CLINICAL TRIAL: NCT05057988
Title: Virtual Empowered Relief for People With Chronic Pain Who Take Methadone or Buprenorphine
Brief Title: Virtual Empowered Relief for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-60855
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: Single intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empowered Relief (Experimental)
  Interventions: Behavioral: Empowered Relief class

INTERVENTIONS:
Behavioral: Empowered Relief class — The participants will attend the Empowered Relief class online via Zoom. The class includes pain neuroscience education, as well as cognition, emotion, and physiologic self-regulation for people with chronic pain. Class participants will learn self-management skills and develop a personalized plan to use the skills every day. Participants will receive an audio file (Relaxation Response) post-class. The class provides patients rapid access to actionable skills for symptom management and pain relief.

SUMMARY:
The purpose of the current pilot study is to examine a feasibility and the preliminary efficacy of Empowered Relief (ER) class when it is delivered 'virtually' to patients with chronic pain who take methadone or buprenorphine. The ER class is a single-session pain management class, which has demonstrated to be effective in improving pain and pain-related distress in patients with chronic low back pain, but its efficacy has not been examined in patients with chronic pain who take methadone or buprenorphine. Class participants will learn self-regulatory skills and develop a personalized plan to use the skills every day. The current study will examine a feasibility and participant's perception and satisfaction of this class at post-class. The study will also follow participants 3 months by administering 5 surveys (baseline, 2 weeks and 1 month, 2 months, and 3 months post-treatment) to determine whether the class confers the short-term and medium-term benefits across various aspects of health.

DETAILED DESCRIPTION:
Some patients with chronic pain are on long-term opioid therapy. Methadone and buprenorphine are often used in long-term opioid therapy for chronic pain. Additionally, chronic pain is highly prevalent in people receiving methadone or buprenorphine for opioid use disorder (MOUD). It is observed that up to 68% of people with MOUD have chronic pain condition. Therefore, a large number of people taking methadone or buprenorphine will suffer from chronic pain, but they frequently face limited availability of clinicians offering non-pharmacological pain management programs. Thus, a brief internet-based pain relief skills program may be one option that can overcome such treatment barrier. A recent randomized control trial on patients with chronic low back pain has demonstrated that a single-session, 2-hour, pain management class (Empowered Relief; ER) was effective to improve pain and pain-related distress. The ER class consists of pain neuroscience education and self-regulatory skills. While the ER is a promising and scalable option, it is not yet tested in patients with chronic pain who take methadone or buprenorphine. The current proposed, single-arm, uncontrolled pilot project will determine a) a feasibility in this patient population, b) patients' perceptions and satisfaction of the ER class and c) preliminary efficacy to inform the design of a future, larger, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Chronic Pain (> 3 months)
* Taking Methadone or Buprenorphine
* English Fluency

Exclusion Criteria:

* Pregnant,
* Gross Cognitive Impairment,
* Acute Suicidality,
* Severe Depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Pain Relief Innovations Lab, Palo Alto, California, United States

REFERENCES:
- [Background] Darnall BD, Roy A, Chen AL, Ziadni MS, Keane RT, You DS, Slater K, Poupore-King H, Mackey I, Kao MC, Cook KF, Lorig K, Zhang D, Hong J, Tian L, Mackey SC. Comparison of a Single-Session Pain Management Skills Intervention With a Single-Session Health Education Intervention and 8 Sessions of Cognitive Behavioral Therapy in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2113401. doi: 10.1001/jamanetworkopen.2021.13401. Erratum In: JAMA Netw Open. 2022 Apr 1;5(4):e229739. doi: 10.1001/jamanetworkopen.2022.9739. PMID 34398206
- [Background] Darnall BD, Sturgeon JA, Kao MC, Hah JM, Mackey SC. From Catastrophizing to Recovery: a pilot study of a single-session treatment for pain catastrophizing. J Pain Res. 2014 Apr 25;7:219-26. doi: 10.2147/JPR.S62329. eCollection 2014. PMID 24851056
- [Background] Ziadni MS, Anderson SR, Gonzalez-Castro L, Darnall BD. Comparative efficacy of a single-session "Empowered Relief" videoconference-delivered group intervention for chronic pain: study protocol for a randomized controlled trial. Trials. 2021 May 22;22(1):358. doi: 10.1186/s13063-021-05303-8. PMID 34022930
- [Background] Klein MR, Darnall BD, You DS. Feasibility of Web-Based Single-Session Empowered Relief in Patients With Chronic Pain Taking Methadone or Buprenorphine: Protocol for a Single-Arm Trial. JMIR Res Protoc. 2024 Jun 6;13:e53784. doi: 10.2196/53784. PMID 38843513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Empowered Relief
Started | 55
Completed | 49
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Empowered Relief
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: missing 2
  Years
    number analyzed (Participants) | 53
    (all) | 49.36 (12.21)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 30
  Male | 22
  Decline/missing | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 40
  More than one race | 2
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Perceived Usefulness
Description: How useful was the information presented in the class? (a single item, 0-10 scale, higher scores correspond to greater perceived usefulness).
Time Frame: once immediately after class
Population: class attenders
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 51
score on a scale | 8.25 (2.34)

2. Primary Outcome: Participant Satisfaction
Description: Please rate your overall satisfaction with the class (a Single Item, 0-10 Scale, higher scores correspond to greater satisfaction).
Time Frame: once immediately after class
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 51
score on a scale | 8.59 (1.96)

3. Primary Outcome: Likelihood of Using the Skills
Description: How likely are you to use the skills and information you learned? (a Single Item, 0-10 Scale, higher scores correspond to greater likelihood)
Time Frame: once immediately after class
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 51
score on a scale | 8.47 (2.14)

4. Secondary Outcome: Pain Bothersomeness
Description: How "bothersome" your pain had been during the previous week? (a Single Item, 0-10 Scale, higher scores greater bothersomeness)
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 50
score on a scale | 5.9 (1.98)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — paired T test; p < .001, t-test, 2 sided; Mean Difference (Net) = 1.04, 95% CI 2-sided [0.53 to 1.55], Standard Deviation 1.80

5. Secondary Outcome: PCS Total Scores
Description: The 13-item Pain Catastrophizing Scale total score ranges from 0 to 52, higher scores correspond to greater pain catastrophizing.
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
score on a scale | 19.02 (11.35)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired T test; p = .208, t-test, 2 sided; Mean Difference (Net) = 0.98, 95% CI 2-sided [-1.42 to 3.37], Standard Deviation 8.17

6. Secondary Outcome: Pain Intensity
Description: How would you rate your pain on average in the past 7 days? (a single item, 0-10 scale, higher scores correspond to greater pain intensity)
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 50
score on a scale | 5.58 (1.70)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired T test; p < .001, t-test, 2 sided; Mean Difference (Net) = 0.86, 95% CI 2-sided [0.52 to 1.20], Standard Deviation 1.20

7. Secondary Outcome: PROMIS-Sleep Disturbance
Description: PROMIS-Sleep Disturbance short form T scores Mean = 50, SD = 10 Higher scores indicate worse symptoms 70T or higher considers severe symptoms
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
T-scores | 57.31 (8.69)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired t test; p = .328, t-test, 1 sided; Mean Difference (Net) = 0.81, 95% CI 2-sided [-.84 to 2.47], Standard Deviation 5.65

8. Other Pre Specified Outcome: PROMIS-Pain Interference
Description: PROMIS-Pain Interference short form T scores Mean = 50, SD = 10 Higher scores indicate worse symptoms 70T or higher considers severe symptoms
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
T-scores | 64.69 (4.89)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired T test; p < .001, t-test, 1 sided; Mean Difference (Final Values) = 2.71, 95% CI 2-sided [1.26 to 4.16], Standard Deviation 4.95

9. Other Pre Specified Outcome: PROMIS-Depression
Description: PROMIS-Depression short form T scores Mean = 50, SD = 10 Higher scores indicate worse symptoms 70T or higher considers severe symptoms
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
T-scores | 57.38 (9.07)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired T test; p = .486, t-test, 1 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-1.22 to 2.53], Standard Deviation 6.38

10. Other Pre Specified Outcome: PROMIS-Anxiety
Description: PROMIS-Anxiety short form T scores Mean = 50, SD = 10 Higher scores indicate worse symptoms 70T or higher considers severe symptoms
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
T-scores | 58.23 (7.96)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired T test; p = .832, t-test, 2 sided; Mean Difference (Final Values) = -.24, 95% CI 2-sided [-2.46 to 1.99], Standard Deviation 7.57

11. Other Pre Specified Outcome: PROMIS-Physical Function
Description: PROMIS-Physical Function short form T Scores Mean = 50, SD = 10 Higher scores indicate better function 30T or higher considers severe impairment
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
T-scores | 35.91 (5.58)
Statistical Analysis 1: Comparison: Empowered Relief; Test type: Other — Paired T test; p = .340, t-test, 2 sided; Mean Difference (Net) = -.43, 95% CI 2-sided [-1.33 to 0.47], Standard Deviation 3.06

12. Other Pre Specified Outcome: Global Impression of Change
Description: The global impression of change (a single item, 1-7 scale, higher scores correspond to greater improvement)
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 49
score on a scale | 4.36 (0.78)

13. Other Pre Specified Outcome: Craving
Description: How much do you crave opiates now? (single item, 0-10 scale, higher scores correspond to greater craving)
Time Frame: At 1 month post-tx
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empowered Relief
Number analyzed (Participants) | 47
score on a scale | 2.43 (2.95)
Statistical Analysis 1: Comparison: Empowered Relief; paired sample t test; Test type: Superiority; p = 0.370, t-test, 2 sided; paired sample t test; Mean Difference (Net) = 0.28, 95% CI 2-sided [-0.34 to 0.89], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Empowered Relief; Test type: Other — Paired T test; p = .370, t-test, 2 sided; Mean Difference (Net) = .28, 95% CI 2-sided [-.34 to .89], Standard Deviation 2.09

ADVERSE EVENTS:
Time Frame: 3 months
Description: None were reported serious adverse events, no one died
Arm/Group | Empowered Relief
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 18/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empowered Relief (N=55)
COVID (Infections and infestations) | 4 (6)
Surgery (Surgical and medical procedures) | 4 (4)
Fall (General disorders) | 4 (4)
Flu/Cold (Infections and infestations) | 3 (3)
Injury/Sprain (Injury, poisoning and procedural complications) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT05057988/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT05057988/SAP_001.pdf